CLINICAL TRIAL: NCT06143449
Title: Taiwan Diabetes Registry (TDR)
Brief Title: Taiwan Diabetes Registry
Status: Recruiting | Type: Observational
Sponsor: The Diabetes Association of the Republic of China (Taiwan) (Other)
Responsible Party: Sponsor
Other Study IDs: Taiwan Diabetes Registry
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study - registry — Observational study - registry

SUMMARY:
To Investigate the Risk Factors, Life Style and Treatments of the Microvascular Disease，Macrovascular Disease and Neuropathy in Patients With Diabetes.

DETAILED DESCRIPTION:
At the first year (2015), the patients ever enrolled into the quality control study by Taiwan Association of Diabetes Educators in 2006 and 2011 will be recruited, and their relevant clinical data will be regularly registered yearly until 2030. In addition, it is planned that type 1 diabetic patients will be enrolled, and their clinical data will be regularly recorded yearly until 2030. Also, newly diagnosed type 2 diabetic patients will be recruited, and their clinical data will be regularly entered to the diabetes web-based system yearly until 2030. We will also include pregnant patients with diabetes since 2023, and their data will be monitored and followed until 2030. Finally, we will also include pregnant patients with diabetes since 2023, and their data will be monitored and followed until 2030.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus

Exclusion Criteria:

* Patients who do not have diabetes mellitus
* Participating in an interventional trial requiring informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Provide data on patient characteristics | Ten years
Provide data on disease management. | Ten years

CONTACTS AND LOCATIONS:
Overall Officials: The Diabetes Association of the Republic of China (Taiwan)
Locations (1):
- The Diabetes Association of the Republic of China (Taiwan), Taipei, Taiwan